CLINICAL TRIAL: NCT02882867
Title: Injuries in Swedish Youth Athletics. The KLUB-study.
Status: Completed | Type: Observational
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Jenny Jacobsson, PhD, PhD, Linkoeping University
Other Study IDs: Dnr 2016/175-31
Record Dates: First submitted 2016-08-22; First posted 2016-08-30 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Athletics Injuries
Keywords: Prospective; Epidemiology; Track and Field
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Injuries in Swedish Youth Athletics. The KLUB-study.

SUMMARY:
It is well known that participation in sports activities as a youth has several health benefits, but at the same time, studies report that the risk is high to obtain injuries related to participation. There is, however, increasing evidence that many of these injuries can be prevented if necessary measures are taken. Prospective studies are therefore needed to be able to plan and carry out measures to prevent the occurrence of injuries. The overall aim of the project KLUB is to study the prevalence and incidence of injuries among athletics youths aged 12-15 years. A particular focus will be placed on identifying factors associated with injury occurrence.

DETAILED DESCRIPTION:
It is well known that participation in sports activities as a youth has several health benefits, but at the same time, studies report that the risk is high to obtain injuries related to participation. There is, however, increasing evidence that many of these injuries can be prevented if necessary measures are taken. So far, most studies examining sports injuries have been conducted on adult elite and among team sports, for example football, ice hockey and bandy. How injury patterns present in individual sports and among youth is not as well documented. A major problem in athletics is that studies have shown an almost identical prevalence and incidence of injury associated with athletics among both young and adult athletes.

Today there are very few published studies on international incidence of injuries among adolescent athletes in athletics and no describing the incidence in Swedish Athletics. These studies have different study design, definitions of injury and rather small groups of athletes, making it difficult to draw conclusions that can be the basis for prevention programs. What after all can be inferred from these previous studies is that injuries related to overuse seems to be most prevalent. Prospective studies are therefore needed to be able to plan and carry out measures to prevent the occurrence of injuries. We intend to carry out an intervention study among athletics youths aged 12-15 years. Before this is carried out, the investigators need to have adequate knowledge of the study population for the effective implementation of the intervention study.

The overall aim of the project KLUB is to study the prevalence and incidence of injuries among athletics youths aged 12-15 years. A particular focus will be placed on identifying factors associated with injury occurrence. The knowledge obtained will be used to allow for injury prevention in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-15 years
* Regularly participate in organized athletics training

Exclusion Criteria:

-

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study is based on a total population design, athletes aged 12-15 years, who regularly participate in organized athletics training in selected clubs (all reachable participants will be invited).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Incidence of injuries in youth athletics | Reporting every second week during one year
  The athletes parents will be asked to provide information regarding training and report any injuries occurring based on the surveillance system developed by Jacobsson et al 2010

SECONDARY OUTCOMES:
Pinpoint risk indicators and factors for different injury types/patterns | Reporting every second week during one year
  The athletes parents will be asked to provide information regarding training and report any injuries occurring based on the surveillance system developed by Jacobsson et al 2010 and Timpka et al 2014

CONTACTS AND LOCATIONS:
Locations (1):
- Swedish Athletics, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jacobsson J, Timpka T, Ekberg J, Kowalski J, Nilsson S, Renstrom P. Design of a protocol for large-scale epidemiological studies in individual sports: the Swedish Athletics injury study. Br J Sports Med. 2010 Dec;44(15):1106-11. doi: 10.1136/bjsm.2009.067678. Epub 2010 May 19. PMID 20484318
- [Background] Timpka T, Alonso JM, Jacobsson J, Junge A, Branco P, Clarsen B, Kowalski J, Mountjoy M, Nilsson S, Pluim B, Renstrom P, Ronsen O, Steffen K, Edouard P. Injury and illness definitions and data collection procedures for use in epidemiological studies in Athletics (track and field): consensus statement. Br J Sports Med. 2014 Apr;48(7):483-90. doi: 10.1136/bjsports-2013-093241. PMID 24620036